CLINICAL TRIAL: NCT03597932
Title: Intraoperative Handover Checklist of Anesthesia Care Improves Postoperative Outcomes Among Patients Undergoing Major Surgery: a Multicenter, Before-after Cohort Study
Brief Title: Intraoperative Handover Checklist of Anesthesia Care Improves Outcomes Among Patients Undergoing Major Surgery
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Collaborators: Zhejiang Provincial Tongde Hospital (Other)
Responsible Party: Principal Investigator, xiangming fang, Director, Head of Anesthesiology and Critical Care, Principal Investigator, Professor, First Affiliated Hospital of Zhejiang University
Other Study IDs: xfang
Record Dates: First submitted 2018-06-22; First posted 2018-07-24 (Actual); Last update posted 2018-07-24 (Actual); Status verified 2018-07

CONDITIONS: Anesthesia; Surgery--Complications; Burnout, Professional
Keywords: major surgery; ansethesia care; postoperative complication; handover checklist; anesthesiologist burnout
MeSH Terms: conditions — Burnout, Professional; Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- baseline or control group: All participant anesthesiologists do intraoperative handover of anesthesia care according to a usual process or without checklist for 2-week to 1-month baseline data collection.
- Checklist group: All participant anesthesiologists do intraoperative handover of anesthesia care by using a standardized handover checklist for another 2-week to 1-month data collection.
  Interventions: Device: standardized handover checklist

INTERVENTIONS:
Device: standardized handover checklist — Following a review of relevant literatures and guidelines, a checklist consisting of the various key items necessary for giving continuing and safe intraoperative patient care was designed and validated by anesthesia residents and staff. Following 2-week to 1-month baseline data collection, each anesthesiologists and anesthesia residents in participating hospitals were asked to implement the safe-anesthesia checklist to improve practice over another 2-week to 1-month period. The checklist consists of an oral confirmation and closed-loop communication between the primary anesthesiologist and the replacement anesthesiologist. Evaluation of the effect of implementation of a standardized checklist during anesthesia care handover on patient safety during follow-up.
  Groups: Checklist group

SUMMARY:
Implementation of a standardized handover checklist for intraoperative anesthesia care transition attenuates burnout among anesthesiologists and improves postoperative outcomes of patients undergoing major surgery , both of which benefit the quality of patient care and the development of anesthesiology.

DETAILED DESCRIPTION:
Many retrospective studies have demonstrated that among adults undergoing major surgery, complete handover of intraoperative anesthesia care compared with no handover was associated with a higher risk of adverse postoperative outcomes. Anesthesiologists keeping on working without handovers may experience symptoms of burnout which do not only pose a threat to the mental and physical health of the anesthesiologist, but also result in sub-optimal safety care of patients. Poor-quality handover without standardized processes can lead to diagnostic and therapeutic delays and precipitate adverse events. An improved system of anesthesia standardized handovers using a checklist would improve transfer of information and professional responsibility and therefore lead to the improvement of patient safety as well as burnout among anesthesiologists. Thus it is urgent to develop a standardized handover checklist for intraoperative anesthesia care to improve postoperative outcome of patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18 years and older undergoing major surgeries requiring a hospital stay of at least 1 night are enrolled in this study.

Exclusion Criteria:

* Adult patients aged less than 18 years undergoing major surgeries and were not requiring a hospital stay of at least 1 night are excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients aged 18 years and older undergoing major surgeries requiring a hospital stay of at least 1 night are enrolled to use a checklist if they need handover of anesthesia care during surgery process.
Sampling Method: Non-Probability Sample
Enrollment: 3342 (Estimated)
Dates: Start 2018-08-01 (Estimated); Primary Completion 2018-08-11 (Estimated); Study Completion 2019-02-28 (Estimated)

PRIMARY OUTCOMES:
Incidence of a composite of all-cause death, hospital readmission, or major postoperative complications | 30 days
  The primary outcome that will be measured is a composite of all-cause death, hospital readmission, or major postoperative complications, all within 30 days post surgery

SECONDARY OUTCOMES:
Incidence of 7 day-, 30 day-, 90 day- and inhospital mortality | 7/30/90 day
  7/30/90-day mortality, inhospital mortality
Incidence of major complications | 30 days
  Postoperative major complications, defined by International Classification of Diseases, Tenth Revision (ICD-10) diagnostic codes
Incidence of ICU admission post surgery | 30 days
  Incidence of postoperative intensive care unit (ICU) admission, ,within 30 days post surgery
The time of hospital length of stay (LOS) | up to 30 days
  Hospital length of stay (LOS)
Incidence of emergency department (ED) visits | 90 days
  Emergency department (ED) visits within 90 days of the index surgery
Any medical cost during hospital stay | up to 90 days
  Any medical cost during hospital stay
Ventilation time within postoperative 30 days | Up to 30 days
  Ventilation time within postoperative 30 days
Anaesthetic resuscitation time | Up to 24 hours
  Anaesthetic resuscitation time after the surgery is completed

CONTACTS AND LOCATIONS:
Overall Officials: Fang Xiangming, Principal Investigator — first affilated hospital of zhejiang university

IPD SHARING:
Plan to Share IPD: Undecided
Share all the data after the first article was published on issue

REFERENCES:
- [Result] Jones PM, Cherry RA, Allen BN, Jenkyn KMB, Shariff SZ, Flier S, Vogt KN, Wijeysundera DN. Association Between Handover of Anesthesia Care and Adverse Postoperative Outcomes Among Patients Undergoing Major Surgery. JAMA. 2018 Jan 9;319(2):143-153. doi: 10.1001/jama.2017.20040. PMID 29318277
- [Result] Li H, Zuo M, Gelb AW, Zhang B, Zhao X, Yao D, Xia D, Huang Y. Chinese Anesthesiologists Have High Burnout and Low Job Satisfaction: A Cross-Sectional Survey. Anesth Analg. 2018 Mar;126(3):1004-1012. doi: 10.1213/ANE.0000000000002776. PMID 29309320
- [Result] van der Wal RA, Bucx MJ, Hendriks JC, Scheffer GJ, Prins JB. Psychological distress, burnout and personality traits in Dutch anaesthesiologists: A survey. Eur J Anaesthesiol. 2016 Mar;33(3):179-86. doi: 10.1097/EJA.0000000000000375. PMID 26575009
- [Result] Segall N, Bonifacio AS, Schroeder RA, Barbeito A, Rogers D, Thornlow DK, Emery J, Kellum S, Wright MC, Mark JB; Durham VA Patient Safety Center of Inquiry. Can we make postoperative patient handovers safer? A systematic review of the literature. Anesth Analg. 2012 Jul;115(1):102-15. doi: 10.1213/ANE.0b013e318253af4b. Epub 2012 Apr 27. PMID 22543067
- [Result] Hudson CC, McDonald B, Hudson JK, Tran D, Boodhwani M. Impact of anesthetic handover on mortality and morbidity in cardiac surgery: a cohort study. J Cardiothorac Vasc Anesth. 2015 Feb;29(1):11-6. doi: 10.1053/j.jvca.2014.05.018. Epub 2014 Nov 24. PMID 25440620
- [Result] Starmer AJ, Spector ND, Srivastava R, West DC, Rosenbluth G, Allen AD, Noble EL, Tse LL, Dalal AK, Keohane CA, Lipsitz SR, Rothschild JM, Wien MF, Yoon CS, Zigmont KR, Wilson KM, O'Toole JK, Solan LG, Aylor M, Bismilla Z, Coffey M, Mahant S, Blankenburg RL, Destino LA, Everhart JL, Patel SJ, Bale JF Jr, Spackman JB, Stevenson AT, Calaman S, Cole FS, Balmer DF, Hepps JH, Lopreiato JO, Yu CE, Sectish TC, Landrigan CP; I-PASS Study Group. Changes in medical errors after implementation of a handoff program. N Engl J Med. 2014 Nov 6;371(19):1803-12. doi: 10.1056/NEJMsa1405556. PMID 25372088
- [Result] Saager L, Hesler BD, You J, Turan A, Mascha EJ, Sessler DI, Kurz A. Intraoperative transitions of anesthesia care and postoperative adverse outcomes. Anesthesiology. 2014 Oct;121(4):695-706. doi: 10.1097/ALN.0000000000000401. PMID 25102312
- [Result] Hyder JA, Bohman JK, Kor DJ, Subramanian A, Bittner EA, Narr BJ, Cima RR, Montori VM. Anesthesia Care Transitions and Risk of Postoperative Complications. Anesth Analg. 2016 Jan;122(1):134-44. doi: 10.1213/ANE.0000000000000692. PMID 25794111
- [Result] Salzwedel C, Bartz HJ, Kuhnelt I, Appel D, Haupt O, Maisch S, Schmidt GN. The effect of a checklist on the quality of post-anaesthesia patient handover: a randomized controlled trial. Int J Qual Health Care. 2013 Apr;25(2):176-81. doi: 10.1093/intqhc/mzt009. Epub 2013 Jan 29. PMID 23360810
- [Result] Lee SC, Atkinson ME, Minard CG, O'Brien A. Electronic tool helps anaesthesia trainee handovers. Clin Teach. 2019 Feb;16(1):58-63. doi: 10.1111/tct.12768. Epub 2018 Mar 6. PMID 29508531
- [Result] Jullia M, Tronet A, Fraumar F, Minville V, Fourcade O, Alacoque X, LeManach Y, Kurrek MM. Training in intraoperative handover and display of a checklist improve communication during transfer of care: An interventional cohort study of anaesthesia residents and nurse anaesthetists. Eur J Anaesthesiol. 2017 Jul;34(7):471-476. doi: 10.1097/EJA.0000000000000636. PMID 28437261